CLINICAL TRIAL: NCT01638039
Title: Identification of Correlates of Protection Against Shigella and Enterotoxigenic Escherichia Coli Infections
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0105-11-HYMC
Record Dates: First submitted 2012-07-08; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Dysentery
MeSH Terms: conditions — Dysentery | interventions — Clinical Laboratory Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diarrheal disease (Active Comparator)
  Interventions: Other: Laboratory Tests
- Control (Active Comparator): Samples of stool, blood, urine saliva
  Interventions: Other: Laboratory Tests

INTERVENTIONS:
Other: Laboratory Tests — Stool, blood, urine and saliva samples

SUMMARY:
The aim of this study is to accelerate the development of vaccine candidates against diarrheal diseases caused by Shigella and Enterotoxigenic Escherichia coli (ETEC). We plan to identify cases of laboratory-proven shigellosis and ETEC-associated diarrhea, to study humoral and cellular immune parameters following natural infections with Shigella and ETEC, and to compare the level of pre-existing local, humoral and cellular immune parameters in cases of shigellosis and ETEC-associated diarrhea and in matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Lab-confirmed Shigella or ETEC
* Individuals or patients without diarrheal disease

Exclusion Criteria:

* n/a

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Identification of cases of shigellosis and ETEC-associated diarrhea | Four years
  Stool of patients examined in laboratory and identified as infected with the pathogens

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cohen, MPH, PhD, Study Director — School of Public Health, Sackler Faculty of Medicine, Tel Aviv University
Locations (7):
- Israel (7):
  - Leumit Health Care System, Petach Tikvah, Elad
  - Emek Medical Center, Afula
  - Hillel Yaffe Medical Center, Hadera
  - Lady Davis Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Sansz Medical Center - Laniado Hospital, Netanya
  - Schneider Children's Medical Center, Petah Tikva